CLINICAL TRIAL: NCT01436825
Title: A Validation Study of the OPTIMS Pharmacokinetic Calculator for Clinician Use in Prophylactic Treatment of Patients With Haemophilia A.
Brief Title: Validation Study of a cOmputer Pharmacokinetic Tool to assIst in the Follow up Care of haeMophilia A Patients
Acronym: OPTIMS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15453; KG110FR (Other: Company internal)
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Haemophilia A
Keywords: Haemophilia A; Factor VIII; Pharmacokinetic; Computer Tool validation
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Prophylactic treatment : 20-40 UI /Kg administered all 2 in 3 days .

SUMMARY:
OPTIMS is a non interventional validation study of the calculator developed by Bayer for clinician's use in the prophylactic treatment by factor VIII of patients with severe or moderate Haemophilia A with a severe clinical profile.

The study takes place during a single visit, at the time of patient enrollment in the study

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe haemophilia A defined as residual factor VIII activity < 1%
* or Patient with moderate haemophilia A (residual factor VIII activity >1% and <5%) with severe clinical profile
* Patient treated in prevention with the same plasma or recombinant factor VIII for at least 6 months
* Patient whose inclusion visit is performed during a routine visit including a measurement of plasma residual factor VIII :c level
* In the medical file (retrospective data) the pharmacokinetic parameters are available and have been obtained from a PK analysis of factor VIII level performed with the same anti haemophilic factor than the one used on the inclusion day

Exclusion Criteria:

* Patients with haemophilia B

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patient with severe haemophilia A defined as residual factor VIII activity < 1%
  * or Patient with moderate haemophilia A (residual factor VIII activity >1% and <5%) with clinical signs of frequent, severe bleeding episodes
  * Patient treated prophylatically with the same plasma or recombinant factor VIII for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The difference of the recovery rate calculated by the physician and the recovery rate calculated by an independent calculator With OPTIMS Tool | after 1 month
The difference of the elimination half-life calculated by the physician and the ones calculated by an independent calculator With OPTIMS Tool | after 1 month
The difference of the clearance calculated by the physician and the ones calculated by an independent calculator With OPTIMS Tool | after 1 month

SECONDARY OUTCOMES:
The dosage of factor VIII calculated by OPTIMS calculator | within 48 hours after enrollment
The practicality of the OPTIMS calculator by a physician's satisfaction questionnaire | within 48 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Many Locations, France
- Many Locations, Italy